CLINICAL TRIAL: NCT05035693
Title: "PMCF MOVE®-C" International, Prospective, Multicentre, Non-randomised Post-market Clinical Follow-up Study Clinical and Radiological Outcome After Mono- and Bisegmental Cervical Intervertebral Disc Prosthetics
Brief Title: Post Market Clinical Follow up Study With the Cervical Disc Prothesis MOVE®-C
Acronym: PMCF_MOVE®-C
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NGMedical GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P004; DRKS00022971 (Other: Deutsches Register Klinischer Studien)
Record Dates: First submitted 2021-03-12; First posted 2021-09-05 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Discopathy; Herniated Cervical Disc; Stenoses, Spinal; Radiculopathy
Keywords: Herniated Disc; Cervical Spine; Discopathy; Radiculopathy
MeSH Terms: conditions — Spinal Stenosis; Radiculopathy; Intervertebral Disc Displacement

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PMCF MOVE-C (Experimental): PMCF MOVE®_C is a single arm observational study with 170 patients.
  Interventions: Device: MOVE®-C

INTERVENTIONS:
Device: MOVE®-C — Momo- or bisegmental implantation of MOVE®-C cervical prothesis.
  Other Names: cervical disc prothesis

SUMMARY:
Study design: International, prospective, multicentre, non-randomised, observational study according to § 23b MPG.

Objectives: Observational study to confirm the safety and performance of the cervical disc prosthesis MOVE®-C.

DETAILED DESCRIPTION:
This clinical investigation is conducted to gain post market results on the Cervical Disc Prosthesis MOVE®-C and to demonstrate the safety and performance. Besides, it is aimed to gain knowledge concerning the development of patients' quality of life (QoL) after the implantation of the Cervical Disc Prosthesis MOVE®-C and to collect data for the analysis of the range of motion (ROM), which is an essential parameter for motion-preserving implants.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of discopathy or disc hernia with radiculopathy or stenosis of the foramen and spinal canal,
2. documented individual history of neck and/or upper extremity pain and/or functional/neurological deficit associated with the cervical level to be treated,
3. no surgical treatment regarding the planned index surgery within the last six weeks prior implantation,
4. unsuccessful conservative medical care regarding the indication within the last six weeks,
5. age ≥18 years,
6. patient must agree to fully participate in the clinical trial and give informed consent in writing,
7. patient is capable to realise the nature, aims and possible consequences of the clinical trial (MPG §20.2.1),
8. patient information has been provided and all written consents of the patient are available.

Exclusion Criteria:

* Known contraindication against the use of cervical intervertebral disc prostheses in accordance with the manufacturer's instructions for use:

  1. Bone mineral density with T-score ≤ -1.5 as determined by spine DXA if male ≥ 60 years of age or female ≥ 50 years of age,
  2. active systemic infection or infection at the operative site,
  3. sustained osteoporotic fracture of the spine, hip or wrist,
  4. spinal metastases,
  5. known allergy to titanium or polycarbonate-urethane,
  6. confirmed pregnancy,
  7. severe cervical myelopathy,
  8. patients requiring a treatment that destabilises the spine (e.g. posterior element decompression),
  9. advanced cervical anatomical deformity at the operative site (e.g. ankylosing spondylitis, scoliosis),
  10. advanced degenerative changes (e.g. spondylosis) at the index vertebral level,
  11. patient is kept in an institution under judicial or official orders (MPG §20.3).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2021-03-11 (Actual); Primary Completion 2025-03-11 (Estimated); Study Completion 2027-03-11 (Estimated)

PRIMARY OUTCOMES:
Improvement from baseline on Neck Disability Index (NDI) | Baseline and month 24
  Primary outcome measure 1 and 2 are combined endpoints. Improvement of the NDI of more than 15 points for a change (pre-postoperative) of up to 30 points with a standard deviation of 25 points.
Improvement from baseline on Visual Analogue Scales (VAS arm/neck) | Baseline and month 24
  Primary outcome measure 1 and 2 are combined endpoints. Improvement of arm and neck pain scale (VAS arm/neck) of more than 2 points at a change (pre-postoperative) of 2.7 points with a standard deviation of 2.5 points.

SECONDARY OUTCOMES:
Change from baseline in Core Outcome Measure Index (COMI neck) | Baseline and months 24
  The clinical results of COMI neck will be compared to the 24 months visit before the operation.
Change from baseline in Short Form 36 Health Survey Questionnaire (SF-36) | Baseline and moths 24
  The clinical results of SF-36 will be compared to the 24 months visit before the operation.
Change from baseline in EuroQoL (EQ-5D-5L) | Baseline and moths 24
  The clinical results of (EQ-5D-5L) will be compared to the 24 months visit before the operation.
Change from baseline in Japanese Orthopedic Association Score (JOA) | Baseline and moths 24
  The clinical results of (JOA) will be compared to the 24 months visit before the operation.
Analyse of the Range of Motion (ROM) | Baseline and moths 24
  The radiological results of the ROM are compared to the 24 months visit before the operation.
Monitoring of product related occurence of adverse events (AE-Monitoring) | Baseline and moths 24
  The radiological results of the AE-Monitoring are compared to the 24 months visit before the operation.

CONTACTS AND LOCATIONS:
Overall Officials: Olaf Süss, PD Dr. med., Principal Investigator — DRK Kliniken Berlin
Locations (7):
- Wiener Gesundheitsverbund-Klinik Penzing, Vienna, Austria
- Germany (6):
  - DRK Klinikum Berlin, Berlin
  - Wirbelsäulenzentrum Fulda Main, Kinzig, Gelnhausen
  - Medizinisches Versorgungszentrum Steinburg, Itzehoe
  - Katholisches Klinikum Koblenz - Montabaur, Koblenz
  - Neurochirurgie am Gasteig, München
  - Rhein-Maas Klinikum Würselen, Würselen

IPD SHARING:
Plan to Share IPD: No
No IPD will be available for other researchers, that will not be a study site in this clinical trial.